CLINICAL TRIAL: NCT06634043
Title: Coronally Advanced Tunnel Combined With Xenogenic Dermal Matrix and L-PRF for the Treatment of Cairo&Amp;#39;s Type 1 and Type 2 Multiple Recessions: A Randomized Comparative Study
Brief Title: Coronally Advanced Tunnel Combined With Xenogenic Dermal Matrix and L-PRF
Acronym: CAF+XADM
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Andres Matteo Pascual La Rocca (Other)
Responsible Party: Sponsor-Investigator, Andres Matteo Pascual La Rocca, DDS, PhD, Alfonso X El Sabio University
Organization: Alfonso X El Sabio University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024 _ 4/269; ORF42414 (Other Grant/Funding Number: Oral Reconstruction Foundation)
Record Dates: First submitted 2024-09-26; First posted 2024-10-09 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Gingival Recession; Gingival Recession, Localized; Mucogingival Defects
Keywords: acellular dermal matrix; coronally advenced tunnel
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: The present study protocol is a two-arm, randomized controlled clinical trial with a follow-up period of 6 months. The protocol of this study has been prepared according to the SPIRIT 2013 Statement. The study will be conducted at the Universidad Alfonso X el Sabio (UAX). Subjects will be recruited consecutively from the Department of Periodontology of Clinica Universitaria de Odontologia (CUO-UAX). The study will be coordinated by the principal investigator. Patients attending the Department of Periodontology (CUO-UAX) will be consecutively screened for eligibility and included in the study by one team member responsible in recruitment .
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization sequence will be carried out using a computer-generated list (StataⓇ v15.1) with a 1:1 allocation ratio according to a block randomization procedure. Allocation concealment will be kept by means of opaque-sealed envelopes that will be opened immediately after the anesthesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Coronally Advanced Tunel + ADM (Novomatrix®)
  Interventions: Procedure: Coronally Advanced Tunel + ADM (Novomatrix®)
- test group (Experimental): Coronally Advanced Tunel + ADM (Novomatrix®) + L-PRF
  Interventions: Procedure: Coronally Advanced Tunel + ADM (Novomatrix®) + L-PRF

INTERVENTIONS:
Procedure: Coronally Advanced Tunel + ADM (Novomatrix®) — ADM (Novomatrix®) will be used alone
  Other Names: Control
  Arms: Control group
Procedure: Coronally Advanced Tunel + ADM (Novomatrix®) + L-PRF — ADM in combination with L-Prf will be applied
  Arms: test group

SUMMARY:
Gingival recession is the exposure of the root surface due to the gum margin moving away from the crown of the tooth. It's common in adults and becomes more prevalent and severe with age. About 50% of people aged 18-64 and up to 88% of those over 65 have at least one site with gingival recession. The causes are multifactorial, including factors like aggressive brushing, thin gum tissue, orthodontic treatments, and more.

A systematic review found that untreated gingival recessions tend to worsen over time, with a significant increase in both the number of sites and the depth of the recession. A new classification system for gingival recessions has been proposed, categorizing them based on the detection of the cementoenamel junction (CEJ) and interproximal attachment loss.

Surgical techniques aim to restore the gum margin to its original position with minimal probing depths and good aesthetic results. The standard treatment involves a connective tissue graft from a donor site, but newer methods using substitutes like collagen matrices and platelet concentrates have shown comparable results.

Acellular Dermal Matrix (ADM) is a processed dermal tissue used as a substitute for connective tissue in root coverage and implant soft tissue corrections. It has shown favorable results, especially in reducing patient morbidity and thickening the gingival phenotype. ADM can be combined with a coronally positioned flap or tunnel technique for effective root coverage.

The use of platelet concentrates, such as Leukocyte and Platelet-Rich Fibrin (L-PRF), has also become an important alternative. These concentrates improve healing by providing growth factors and cytokines, aiding in the development of microvascularization.

The objective is to assess whether combining Acellular Dermal Matrix (ADM) with Leukocyte and Platelet-Rich Fibrin (L-PRF) yields better or comparable results to ADM alone in terms of complete root coverage, percentage of root coverage (PRC), recession reduction (RecRED), gain of keratinized gingiva (KGG), height of the interdental papilla (IDH), and increased gingival thickness (GT) after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with ≥18 years of age. ability to understand all the study procedures and to comply with them throughout the entire study period. Ability and willingness to give written informed consent.

an adequate level of oral hygiene (plaque index ≤ 25%) (O'Leary et al., 1972).

an adequate general bleeding on probing (≤ 20%) treated periodontal disease. presence of two or more adjacent Cairo type I or II gingival recessions, with ≥1mm of keratinized gingiva in all the deffects.

Exclusion Criteria:

* untreated periodontitis.
* smokers > 5 cigarettes per day.
* local or systemic diseases that would interfere with routine periodontal therapy (i.e., uncontrolled diabetes mellitus, cancer, HIV, chronic high-dose steroid therapy, metabolic bone disease, radiation, immunosuppressive disease, hepatic dysfunction, immunosuppressive disease, autoimmune disease).
* treatment with anticoagulants or bisphosphonates.
* pregnant or lactating women.
* radiographic interproximal bone loss.
* tooth Mobility. If present, splinting should be performed prior to treatment.
* Active orthodontic treatment
* allergy or intolerance to study medication
* use of systemic antibiotics during the last 3 months
* use of systemic antibiotics for endocarditis prophylaxis
* patients with intentions to change residence that prevent follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Root Coverage | 6 months
  Percentage of root coverage after 6 month

SECONDARY OUTCOMES:
Patients satisfaction | 6 months
  health-related quality-of-life tool,specified on root coverage procedures, with a 0 to 10 pointscale used for assessing the level of concern of the following patient-centered criteria: a) general esthetics, b)cost/benefit c)general experience.
  10 being the best and 0 being the poorest score.
Patients Morbidity | 6 months
  Post Operative pain measured with visual analogue scale where the level of pain will be assessed according to the grades from 0 to 10.
presence of dentin hipersensitivity | 6 months
  Measured with a visual analogue scale after external stimuli applied to the surface of exposed dentin with open tubules, the level of pain will be assessed according to the grades of pain from 0 to 10.
Pink Esthetic Scores results | 6 months
  The pink esthetic score (PES) provides a reproducible method for evaluating papilla form as well as other soft tissue variables including color and surface.
  The PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft-tissue contour, alveolar process deficiency, soft-tissue color and texture.
  Each variable will be assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score.
presence of dentin hipersensitivity | 6 months
  Measured with a visual analogue scale after external stimuli applied to the surface of exposed dentin with open tubules, he level of pain will be assessed according to the grades of pain from 0 to 10.

IPD SHARING:
Plan to Share IPD: Undecided